CLINICAL TRIAL: NCT04372017
Title: Randomized, Double-Blind, Controlled Trial of Hydroxychloroquine vs Placebo as Post-Exposure Prophylaxis Against COVID-19 Infection
Brief Title: Hydroxychloroquine as Post-Exposure Prophylaxis Against COVID-19 Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unlikelihood of benefit based on other studies.
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PEPCOH
Record Dates: First submitted 2020-04-25; First posted 2020-05-01 (Actual); Results first posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; SARS-CoV 2
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A: Healthcare worker (hydroxychloroquine) (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Cohort A: Healthcare worker (placebo) (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D
- Cohort B: High-Risk participant (hydroxychloroqine) (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Cohort B: High-Risk participant (placebo) (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Hydroxychloroquine — Participants randomized to hydroxychloroquine will take 800mg on day 1 followed by 400mg on days 2-5.
  Arms: Cohort A: Healthcare worker (hydroxychloroquine); Cohort B: High-Risk participant (hydroxychloroqine)
Dietary Supplement: Vitamin D — Participants randomized to placebo will take IU1600 on day 1 and IU 800 on days 2-5.
  Arms: Cohort A: Healthcare worker (placebo); Cohort B: High-Risk participant (placebo)

SUMMARY:
This is a prospective, double-blind, randomized, placebo-controlled study in two distinct cohorts to evaluate the efficacy and safety of hydroxychloroquine in the prevention of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Cohort A:

* ≥ 18 years old
* Employee of healthcare organization in South Dakota or Sanford Health employee in any location and with exposure to a person with COVID-19 within the last 5 days

  * Occupational exposure as determined by the participant's employee health department (i.e. not wearing the proper Personal Protective Equipment (PPE))
  * Criteria according to Center for Disease Control (CDC) guidelines
  * Community exposure (within 6 feet for at least 15 minutes)
* No current symptoms attributable to COVID-19, per HCW report (fever, cough, difficulty breathing, sore throat)
* No prior COVID-19 positive diagnosis (eligible if previous testing is negative and meets all other inclusion and exclusion)
* Ability to provide informed consent

Inclusion Criteria - Cohort B

* ≥ 18 years old
* High-risk person who had close contact (i.e. within 6 feet for at least 15 minutes) with a COVID-19 positive person within the last 5 days and is a South Dakota resident or high-risk person with close household contact of a COVID-19 positive Sanford employee
* High-risk person defined by:
* Age 18-44 with 2 or more comorbidities listed below
* Age 45-79 with any comorbid condition listed below
* Age 80 and above (regardless of comorbid conditions)
* Co-morbid list

  * Congestive Heart Failure (CHF)
  * Chronic lung disease (Includes any of the following: asthma, chronic obstructive pulmonary disease, emphysema)
  * Solid organ transplant or immunosuppression (Defined as an outpatient prescription of greater than 10 mg/day of prednisone or equivalent, use of chemotherapy, or use of immunosuppressive agents for solid organ transplant or for an autoimmune disease.)
  * Chronic Kidney Disease or End Stage Renal Disease
  * Diabetes mellitus
  * Cardiovascular disease/Hypertension
  * Smoking/Vaping (currently using or history of using in the past 1 year)
  * Obesity (calculated by height and weight per participant report)
  * Hyperlipidemia
* No current symptoms attributable to COVID-19
* No prior COVID-19 positive diagnosis (eligible if previous testing is negative and meets all other inclusion and exclusion)
* Ability to provide informed consent
* Confirmed review of concomitant medications (with emphasis on cardiac medications)

Exclusion Criteria Cohort A & B:

* Known allergy to hydroxychloroquine or quinine
* Known history of long QT syndrome
* Known history of arrhythmia or dysrhythmia
* Known current QTc >500 ms
* Known G6PD deficiency
* Known history of hypoglycemia
* Pregnant or Nursing by patient history
* Use of any of the following concomitant medications: See Appendix D for Exclusion medication list
* Concurrent diagnosis of dermatitis, porphyria, or psoriasis
* History of chronic liver disease, including cirrhosis and/or diagnosis of hepatitis (infectious, idiopathic, or immune)
* History of chronic kidney disease
* Pre-existing retinopathy
* Already taking hydroxychloroquine
* Any condition or medication in the opinion of the investigator that would prohibit the use of hydroxychloroquine
* Enrollment in another clinical with investigational drug or device
* Inability to swallow pills
* Adults unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hoover, MD, Study Chair — Sanford Health
Locations (1):
- Sanford Health, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A: Healthcare Worker (Hydroxychloroquine) | Cohort A: Healthcare Worker (Placebo) | Cohort B: High-Risk Participant (Hydroxychloroqine) | Cohort B: High-Risk Participant (Placebo)
Started | 1 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects or data analyzed. Study was closed to enrollment before analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Healthcare Worker (Hydroxychloroquine) | Cohort A: Healthcare Worker (Placebo) | Cohort B: High-Risk Participant (Hydroxychloroqine) | Cohort B: High-Risk Participant (Placebo) | Total
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  |  | 0
  Between 18 and 65 years | 1 |  |  |  | 1
  >=65 years | 0 |  |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  |  |  | 0
  Male | 1 |  |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  |  | 0
  Not Hispanic or Latino | 0 |  |  |  | 0
  Unknown or Not Reported | 1 |  |  |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  | 0
  Asian | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  | 0
  Black or African American | 0 |  |  |  | 0
  White | 0 |  |  |  | 0
  More than one race | 0 |  |  |  | 0
  Unknown or Not Reported | 1 |  |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Percentage of COVID-19 Exposed Healthcare Workers Treated With Hydroxychloroquine With a Positive COVID-19 Test.
Description: Determine whether post-exposure prophylaxis with hydroxychloroquine can prevent COVID-19 in healthcare workers who have been exposed to a known case of COVID-19.
Time Frame: At enrollment completion outcome 1 will be analyzed.
Population: No subject data was analyzed. Study was closed early.
Arm/Group | Cohort A: Healthcare Worker (Hydroxychloroquine) | Cohort A: Healthcare Worker (Placebo) | Cohort B: High-Risk Participant (Hydroxychloroqine) | Cohort B: High-Risk Participant (Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Cohort B: Percentage of COVID-19 Exposed High-risk Individuals Treated With Hydroxychloroquine With a Positive COVID-19 Test.
Description: Determine whether post-exposure prophylaxis with hydroxychloroquine can prevent COVID-19 in high-risk individuals who have been exposed to a known case of COVID-19.
Time Frame: At enrollment completion outcome 2 will be analyzed.
Population: No subject data was analyzed. Study was closed early.
Arm/Group | Cohort A: Healthcare Worker (Hydroxychloroquine) | Cohort A: Healthcare Worker (Placebo) | Cohort B: High-Risk Participant (Hydroxychloroqine) | Cohort B: High-Risk Participant (Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 of treatment through 12 months after day 1.
Description: No enrollments to Cohort B. No enrollments to Cohort A (Healthcare Worker-Placebo).
  CT CAE criteria was used for the 1 participant on Cohort A (Healthcare Worker-Hydroxychloroquine)
Arm/Group | Cohort A: Healthcare Worker (Hydroxychloroquine) | Cohort A: Healthcare Worker (Placebo) | Cohort B: High-Risk Participant (Hydroxychloroqine) | Cohort B: High-Risk Participant (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Healthcare Worker (Hydroxychloroquine) (N=1) | Cohort A: Healthcare Worker (Placebo) (N=0) | Cohort B: High-Risk Participant (Hydroxychloroqine) (N=0) | Cohort B: High-Risk Participant (Placebo) (N=0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Covid-19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT04372017/Prot_SAP_002.pdf
  • Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT04372017/ICF_003.pdf